CLINICAL TRIAL: NCT01839331
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy and Safety of Two Doses of Intra-Articular Injection of Ampion™ in Adults With Pain Due to Osteoarthritis of the Knee
Brief Title: An Efficacy and Safety Study of Two Doses of Intra-Articular Ampion Injection for Pain of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-003-A
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ampion 4 mL Dose (Experimental): 4 mL Injection of Ampion
  Interventions: Biological: 4 mL injection of Ampion
- Placebo 4 mL Dose (Placebo Comparator): 4 mL Injection of Placebo
  Interventions: Drug: 4 mL Injection of Placebo
- Ampion 10 mL Dose (Experimental): 10 mL Injection of Ampion
  Interventions: Biological: 10 mL Injection of Ampion
- Placebo 10 mL Dose (Placebo Comparator): 10 mL Injection of Placebo
  Interventions: Drug: 10 mL Injection of Placebo

INTERVENTIONS:
Biological: 4 mL injection of Ampion — 4 mL Injection of Ampion
  Arms: Ampion 4 mL Dose
Biological: 10 mL Injection of Ampion — 10 mL Injection of Ampion
  Arms: Ampion 10 mL Dose
Drug: 4 mL Injection of Placebo — 4 mL Injection of Placebo
  Other Names: Saline
  Arms: Placebo 4 mL Dose
Drug: 10 mL Injection of Placebo — 10 mL Injection of Placebo
  Other Names: Saline
  Arms: Placebo 10 mL Dose

SUMMARY:
This study will evaluate the efficacy of two doses of Intra-Articular Injection of Ampion™ in Adults with pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
A Randomized, Placebo-controlled, Double-Blind Study to Evaluate the Efficacy and Safety of two Doses of Intra-Articular Injection of Ampion™ in Adults with pain due to osteoarthritis of the knee.

The primary trial objective is to evaluate whether there is greater efficacy of 10 mL Ampion™ versus 10 mL placebo than 4 mL Ampion™ versus 4 mL placebo intra-articular (IA) injection in improving knee pain, when applied to patients suffering from OA of the knee.

The secondary trial objective include: the evaluation of the safety of an intra-articular injection of Ampion™ when applied to patients suffering from OA of the knee, evaluation of the efficacy of intra-articular injection of Ampion™ and placebo on stiffness and function when applied to patients suffering from OA of the knee and evaluation of responder status defined by the Outcome Measures in Rheumatology Clinical Trials and Osteoarthritis Research Society International (OMERACT-OARSI) Criteria.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate in the study
* Willing and able to comply with all study requirements and instructions of the site study staff
* Male or female, 40 years to 85 years old (inclusive)
* Must be ambulatory
* Index knee must be symptomatic for greater than 6 months with a clinical diagnosis of osteoarthritis (OA) and supported by radiological evidence Kellgren Lawrence Grade II to IV) that is not older than 6 months prior to the date of screening
* Moderate to moderately-severe OA pain in the index knee (rating of at least 1.5 on the WOMAC Index 3.1 5-point Likert Pain Subscale) assessed at screening
* Moderate to moderately-severe OA pain in the index knee (even if chronic doses of nonsteroidal anti-inflammatory drug (NSAID), which have not changed in the 4 weeks prior to screening, have been/are being used)
* No analgesia (including acetaminophen [paracetamol]) taken 12 hours prior to an efficacy measure
* No known clinically significant liver abnormality e.g. cirrhosis, transplant, etc.)

Exclusion Criteria:

* As a result of medical review and screening investigation, the Principal Investigator considers the patient unfit for the study
* A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion)
* A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate)
* Presence of tense effusions
* Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the affected knee, as assessed locally by the Principal Investigator
* Isolated patella femoral syndrome, also known as chondromalacia
* Any other disease or condition interfering with the free use and evaluation of the index knee for the duration of the trial e.g. cancer, congenital defects, spine OA)
* Major injury to the index knee within the 12 months prior to screening
* Severe hip OA ipsilateral to the index knee
* Any pain that could interfere with the assessment of index knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee)
* Any pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study
* Use of the following medications:

  1. No IA injected pain medications in the study knee during the study
  2. No analgesics containing opioids. NSAIDs may be continued at levels preceding the study and acetaminophen is available as a rescue medication during the study from the provided supply
  3. No topical treatment on osteoarthritis index knee during the study
  4. No significant anticoagulant therapy (e.g. Heparin or Lovenox) during the study (treatment such as Aspirin and Plavix are allowed)
  5. No systemic treatments that may interfere with safety or efficacy assessments during the study
  6. No immunosuppressants
  7. No use of corticosteroids > 10 mg prednisolone equivalent per day (if ≤ 10 mg prednisolone, the dose must be stable)
* Any human albumin treatment in the 3 months before randomization

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2013-08-19 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, Study Director — Ampio Pharmaceuticals. Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bar-Or D, Salottolo KM, Loose H, Phillips MJ, McGrath B, Wei N, Borders JL, Ervin JE, Kivitz A, Hermann M, Shlotzhauer T, Churchill M, Slappey D, Clift V. A randomized clinical trial to evaluate two doses of an intra-articular injection of LMWF-5A in adults with pain due to osteoarthritis of the knee. PLoS One. 2014 Feb 3;9(2):e87910. doi: 10.1371/journal.pone.0087910. eCollection 2014. PMID 24498399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects occurred in medical clinics during the months of March, April, and May 2013.
Pre-assignment Details: No pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study.
Units Other Than Participants: Single knee
Period: Overall Study
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose | Ampion 10 mL Dose | Placebo 10 mL Dose
Started | 83; 83 Single knee | 83; 83 Single knee | 82; 82 Single knee | 81; 81 Single knee
Week 6 | 83; 83 Single knee | 83; 83 Single knee | 82; 82 Single knee | 81; 81 Single knee
Completed | 79; 79 Single knee | 77; 77 Single knee | 77; 77 Single knee | 76; 76 Single knee
Not Completed | 4; 4 Single knee | 6; 6 Single knee | 5; 5 Single knee | 5; 5 Single knee
Not completed — Early Termination | 3 | 0 | 1 | 2
Not completed — Protocol Violation | 1 | 6 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose | Ampion 10 mL Dose | Placebo 10 mL Dose | Total
Number analyzed (Participants) | 83 | 83 | 82 | 81 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.27) | 60.7 (8.27) | 62.8 (8.36) | 63.8 (9.95) | 62.48 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 57 | 46 | 50 | 209
  Male | 27 | 26 | 36 | 31 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 83 | 83 | 80 | 79 | 325
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 8 | 8 | 4 | 29
  White | 74 | 74 | 74 | 77 | 299
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 83 | 82 | 81 | 329
Weight (kg) [Mean (Standard Deviation); unit: kg] | 95.6 (22.15) | 98.4 (25.28) | 95.2 (22.42) | 90.6 (22.07) | 94.98 (23.08)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 33.2 (7.76) | 34.5 (8.02) | 32.8 (6.58) | 32.1 (6.46) | 33.16 (7.27)
Kellgren-Lawrence (KL) Grade [Count of Participants; unit: Participants] — Kellgren-Lawrence grading is based on the radiologic features of osteoarthritis.
  Ann Rheum Dis. 1957;16:494-502.
  Grade II (Mild): Definite osteophytes, possible joint space narrowing. Grade III (Moderate): Moderate osteophytes, definite joint space narrowing, some sclerosis, possible bone-end deformity.
  Grade IV (Severe): Large osteophytes, marked joint space narrowing, severe sclerosis, definite bone ends deformity.
  Participants
    Kellgren-Lawrence Grade II | 28 | 29 | 32 | 26 | 115
    Kellgren-Lawrence Grade III | 38 | 32 | 35 | 34 | 139
    Kellgren-Lawrence Grade IV | 17 | 22 | 15 | 21 | 75
WOMAC Pain [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Pain Score.
  Higher scores are indicative of higher levels of self-reported pain.
  score on a scale | 2.22 (0.490) | 2.32 (0.548) | 2.19 (0.512) | 2.23 (0.602) | 2.24 (0.54)
WOMAC Stiffness [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates stiffness (2 items): after first waking and later in the day.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Stiffness Score.
  Higher scores are indicative of higher levels of self-reported joint stiffness.
  score on a scale | 2.25 (0.717) | 2.36 (0.798) | 2.43 (0.781) | 2.44 (0.768) | 2.37 (0.77)
WOMAC Function [Mean (Standard Deviation); unit: score on a scale] — WOMAC 3.1 evaluates Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy/light domestic duties.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 17 scores constitutes the Baseline Function Score.
  Higher scores are indicative of higher levels of limitations of self-reported physical function.
  score on a scale | 2.13 (0.564) | 2.25 (0.626) | 2.23 (0.610) | 2.22 (0.616) | 2.21 (0.60)
Patient's Global Assessment (PGA) [Mean (Standard Deviation); unit: score on a scale] — The Patient's Global Assessment of disease severity has subjects answer the following question: "Considering all the ways in which your arthritis affects you, please indicate how you are doing." Patients respond by using a 5-point Likert score (0=very well; 1=well; 2=fair; 3=poor; 4=very poor).
  Higher scores indicate greater patient's assessment of disease severity due to arthritis.
  score on a scale | 3.35 (0.652) | 3.40 (0.811) | 3.35 (0.822) | 3.42 (0.652) | 3.38 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Pain
Description: Mean Change in WOMAC A Pain (Western Ontario and McMaster Universities Arthritis Index) score from Baseline to 12 weeks. 5-point Likert scale (0=none to 4=extreme). A negative difference constitutes a decrease in pain with a greater negative value indicating a greater reduction in pain.
Time Frame: Scored at Baseline and 12 weeks
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Ampion Combined (4 mL & 10 mL Dose): Combined results of 4 mL and 10 mL Ampion dose
- Placebo Combined (4 mL and 10 mL Dose): Combined results of 4 mL and 10 mL Placebo dose
Arm/Group | Ampion Combined (4 mL & 10 mL Dose) | Placebo Combined (4 mL and 10 mL Dose) | Ampion 4 mL Dose | Placebo 4 mL Dose | Ampion 10 mL Dose | Placebo 10 mL Dose
Number analyzed (Participants) | 165 | 164 | 83 | 83 | 82 | 81
score on a scale | -0.93 [-1.045 to -0.807] | -0.72 [-0.852 to -0.587] | -0.93 [-1.099 to -0.766] | -0.71 [-0.871 to -0.543] | -0.92 [-1.093 to -0.746] | -0.73 [-0.946 to -0.520]
Statistical Analysis 1: Comparison: Ampion Combined (4 mL & 10 mL Dose) vs Placebo Combined (4 mL and 10 mL Dose); Test type: Superiority; p = 0.004, ANOVA — Adjusted for injection volume (4 mL or 10 mL) and baseline WOMAC score
Statistical Analysis 2: Comparison: Ampion 4 mL Dose vs Placebo 4 mL Dose; Test type: Superiority; p = 0.017, ANOVA — Adjusted for injection volume and baseline WOMAC score
Statistical Analysis 3: Comparison: Ampion 10 mL Dose vs Placebo 10 mL Dose; Test type: Superiority; p = 0.093, ANOVA — Adjusted for injection volume and baseline WOMAC score

2. Secondary Outcome: Change in Knee Function
Description: Mean change in WOMAC C function score (Western Ontario and McMaster Universities Arthritis Index) from Baseline to 12 weeks. 5-point Likert scale indicating limitation of function (0=none to 4=extreme). A greater negative value indicates a improvement in function.
Time Frame: Scored at Baseline and 12 weeks.
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Ampion Combined (4 mL and 10 mL) Dose: Combined results of 4 mL and 10 mL Ampion Dose
- Placebo Combined (4 mL and 10 mL) Dose: Combined results of 4 mL and 10 mL Placebo dose results
Arm/Group | Ampion Combined (4 mL and 10 mL) Dose | Placebo Combined (4 mL and 10 mL) Dose | Ampion 4 mL Dose | Placebo 4 mL Dose | Ampion 10 mL Dose | Placebo 10 mL Dose
Number analyzed (Participants) | 165 | 164 | 83 | 83 | 82 | 81
score on a scale | -0.78 [-0.901 to -0.655] | -0.64 [-0.766 to -0.510] | -0.72 [-0.899 to -0.549] | -0.58 [-0.735 to -0.429] | -0.83 [-1.007 to -0.657] | -0.69 [-0.903 to -0.485]
Statistical Analysis 1: Comparison: Ampion Combined (4 mL and 10 mL) Dose vs Placebo Combined (4 mL and 10 mL) Dose; Test type: Superiority — Adjusted for injection volume (4 mL or 10 mL) and baseline WOMAC score; p = 0.0442, ANOVA

3. Secondary Outcome: Change in Knee Stiffness.
Description: Mean Change in WOMAC B stiffness score from Baseline to 12 weeks. 5-point Likert scale (0=none to 4=extreme). A negative difference constitutes a reduction in stiffness.
Time Frame: Scored at Baseline and 12 weeks.
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo Combined (4 mL and 10 mL) Dose: Combined results of 4 mL and 10 mL Placebo dose
Arm/Group | Ampion Combined (4 mL and 10 mL) Dose | Placebo Combined (4 mL and 10 mL) Dose | Ampion 4 mL Dose | Placebo 4 mL Dose | Ampion 10 mL Dose | Placebo 10 mL Dose
Number analyzed (Participants) | 165 | 164 | 83 | 83 | 82 | 81
score on a scale | -0.72 [-0.866 to -0.582] | -0.67 [-0.823 to -0.524] | -0.66 [-0.860 to -0.465] | -0.55 [-0.746 to -0.350] | -0.79 [-0.994 to -0.579] | -0.80 [-1.028 to -0.577]
Statistical Analysis 1: Comparison: Ampion Combined (4 mL and 10 mL) Dose vs Placebo Combined (4 mL and 10 mL) Dose; Test type: Superiority; p = 0.4133, ANOVA — Adjusted for injection volume (4 mL or 10 mL) and baseline WOMAC score

4. Secondary Outcome: Change in Patient's Global Assessment
Description: Patients are asked the following question: "Considering all the ways in which your arthritis affects you, please indicate how you are doing." 5-point Likert scale (0 = very well, 1 = well, 2 = fair, 3 = poor, 4 = very poor). A negative value constitutes an improvement in patient's assessment of disease severity.
Time Frame: Scored at Baseline and 12 weeks.
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ampion Combined (4 mL and 10 mL) Dose | Placebo Combined (4 mL and 10 mL) Dose | Ampion 4 mL Dose | Placebo 4 mL Dose | Ampion 10 mL Dose | Placebo 10 mL Dose
Number analyzed (Participants) | 165 | 164 | 83 | 83 | 82 | 81
score on a scale | -0.87 [-1.033 to -0.701] | -0.65 [-0.821 to -0.472] | -0.96 [-1.186 to -0.742] | -0.55 [-0.801 to -0.308] | -0.77 [-1.018 to -0.519] | -0.74 [-0.992 to -0.489]
Statistical Analysis 1: Comparison: Ampion Combined (4 mL and 10 mL) Dose vs Placebo Combined (4 mL and 10 mL) Dose; Test type: Superiority; p = 0.0122, ANOVA — Adjusted for injection volume (4 mL or 10 mL) and baseline PGA

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Patients will be followed for the occurrence of Adverse Events (AEs) until 12 weeks after the first dose of study medication and additionally for AEs in the study knee for those patients who opt to continue in the 20 week follow-up visit.
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose | Ampion 10 mL Dose | Placebo 10 mL Dose
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/83 | 0/82 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/83 | 2/83 | 3/82 | 2/81
Other Adverse Events (participants affected / at risk) | 23/83 | 38/83 | 17/82 | 29/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampion 4 mL Dose (N=83) | Placebo 4 mL Dose (N=83) | Ampion 10 mL Dose (N=82) | Placebo 10 mL Dose (N=81)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampion 4 mL Dose (N=83) | Placebo 4 mL Dose (N=83) | Ampion 10 mL Dose (N=82) | Placebo 10 mL Dose (N=81)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 16 (16) | 6 (6) | 8 (8)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Injection Site Pain (General disorders) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Ligament Sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The relatively small number of subjects in each arm may account for lack of statistical significance of improvement in Knee pain of 10 mL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less